CLINICAL TRIAL: NCT04368390
Title: Imaging Analysis of COVID-19 + Patients With Abnormal Neurological Examination
Brief Title: Neuroradiolological Analysis of COVID-19 Patients
Acronym: NEURO-COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7759
Record Dates: First submitted 2020-04-28; First posted 2020-04-29 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-04

CONDITIONS: Covid-19
Keywords: COVID-19; MRI; Brain
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To describe the radiological presentation of brain abnormalities in COVID-19 + patients

ELIGIBILITY:
Inclusion Criteria:

* Adults
* COVID-19 +
* Abnormal neurological examination
* who underwent a brain MRI

Exclusion Criteria:

* No participation agreement
* Non COVID-19 patients
* Patients COVID-19 + without neurological abnormality or without MRI examination

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients COVID-19 with abnormal neurological examination
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-04-03 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Neuroradiological analysis of patients brain MRI | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Imagerie 2 - Neuroradiologie, Strasbourg, France

REFERENCES:
- [Derived] Kremer S, Lersy F, Anheim M, Merdji H, Schenck M, Oesterle H, Bolognini F, Messie J, Khalil A, Gaudemer A, Carre S, Alleg M, Lecocq C, Schmitt E, Anxionnat R, Zhu F, Jager L, Nesser P, Mba YT, Hmeydia G, Benzakoun J, Oppenheim C, Ferre JC, Maamar A, Carsin-Nicol B, Comby PO, Ricolfi F, Thouant P, Boutet C, Fabre X, Forestier G, de Beaurepaire I, Bornet G, Desal H, Boulouis G, Berge J, Kazemi A, Pyatigorskaya N, Lecler A, Saleme S, Edjlali-Goujon M, Kerleroux B, Constans JM, Zorn PE, Mathieu M, Baloglu S, Ardellier FD, Willaume T, Brisset JC, Caillard S, Collange O, Mertes PM, Schneider F, Fafi-Kremer S, Ohana M, Meziani F, Meyer N, Helms J, Cotton F. Neurologic and neuroimaging findings in patients with COVID-19: A retrospective multicenter study. Neurology. 2020 Sep 29;95(13):e1868-e1882. doi: 10.1212/WNL.0000000000010112. Epub 2020 Jul 17. PMID 32680942